CLINICAL TRIAL: NCT07275684
Title: Antimicrobial Efficacy of Charcoal-impregnated Toothbrushes: a Randomized Controlled Clinical Study.
Brief Title: Charcoal Toothbrushes and Bacterial Contamination: a Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed V University in Rabat (Other)
Collaborators: Oral Biotechnology Laboratory, Faculty of Dental Medicine, Mohammed V University in Rabat (Unknown)
Responsible Party: Principal Investigator, Asmae Digoug, Specialist in Conservative Dentistry, Faculty of Dental Medicine Rabat, Mohammed V University in Rabat
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CERB 44-25
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Oral Hygiene; Toothbrush Contamination; Bacterial Contamination
Keywords: Charcoal toothbrush; Oral hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Charcoal-Impregnated Toothbrush (Experimental): Participants use a Colgate Double Action Medium toothbrush with charcoal-impregnated bristles twice daily for 2 minutes using the rolling technique. They use standardized fluoride toothpaste (1450 ppm) and follow instructions for proper storage: vertical position, bristles up, uncovered, at least 1-2 meters from toilets. Participants record their daily brushing in a standardized log sheet.
  Interventions: Device: Charcoal-Impregnated Toothbrush
- Conventional Toothbrush (Active Comparator): Participants use a Colgate Double Action Medium toothbrush without charcoal twice daily for 2 minutes using the rolling technique. They use the same standardized fluoride toothpaste (1450 ppm) and follow the same storage and logging instructions as Arm 1.
  Interventions: Device: Conventional Toothbrush

INTERVENTIONS:
Device: Charcoal-Impregnated Toothbrush — Participants use the Colgate Double Action Medium toothbrush with charcoal bristles as described in Arm 1. Daily brushing is twice for 2 minutes, using the rolling technique, with standardized fluoride toothpaste (1450 ppm). Proper storage instructions and daily log recording are followed.
  Arms: Charcoal-Impregnated Toothbrush
Device: Conventional Toothbrush — Participants use the Colgate Double Action Medium toothbrush without charcoal bristles as described in Arm 2. Daily brushing is twice for 2 minutes, using the rolling technique, with standardized fluoride toothpaste (1450 ppm). Proper storage instructions and daily log recording are followed.
  Arms: Conventional Toothbrush

SUMMARY:
This randomized controlled clinical trial aims to evaluate the antibacterial effectiveness of toothbrushes with charcoal-impregnated bristles compared to conventional toothbrushes without charcoal. The main objective is to assess and compare the microbial contamination on the toothbrushes after 21 days of use.

Thirty-two healthy dental students from the Faculty of Dental Medicine of Rabat (16 males and 16 females, aged 18-24) were enrolled through convenience sampling. Participants were randomly assigned to two groups:

Group A: Colgate Double Action Medium toothbrushes with charcoal-impregnated bristles.

Group B: Colgate Double Action Medium toothbrushes without charcoal (control group).

Participants brushed their teeth twice daily for two minutes using the rolling technique and a standardized fluoride toothpaste (1450 ppm). They were instructed not to use mouthwash or antiseptic toothpaste, to rinse brushes only with tap water (without touching the bristles), to store them vertically with bristles facing upward, and to keep them uncovered and at least one meter away from toilets.

After 21 days, used toothbrushes were collected in sterile pouches and transferred to the microbiology laboratory. A quarter of the bristles from each brush head was aseptically cut, immersed in sterile saline solution, and vortexed to dislodge microorganisms. Aliquots of 200 µL were inoculated onto blood agar (Columbia agar base enriched with sterile blood). After incubation at 37°C for 48 hours, colony-forming units (CFU) were manually counted to estimate microbial contamination levels (CFU/mL).

Clinical data (Silness and Löe plaque index, Löe and Silness gingival index, and DMF index) were collected at baseline.

Statistical analysis was performed using Jamovi software. The comparison of CFU counts between groups aimed to determine whether charcoal impregnation reduces microbial contamination of toothbrush bristles.

This study involves minimal risk and no investigational drug or device. Ethical approval was obtained from the Ethics Committee of the Faculty of Dental Medicine of Rabat.

DETAILED DESCRIPTION:
1. Background and Rationale

   Toothbrushes are essential oral hygiene tools, but they can act as reservoirs for microorganisms due to their humid storage environment. This bacterial colonization may reintroduce pathogens into the oral cavity, increasing the risk of oral and systemic infections. Activated charcoal, known for its adsorption capacity and antibacterial potential, has been incorporated into dental products, including toothbrush bristles. However, evidence regarding its effect on bacterial contamination of toothbrushes remains limited.

   This trial aims to evaluate whether charcoal-infused bristles reduce microbial contamination compared to standard nylon bristles after 21 days of regular use.
2. Study Objectives

   Primary Objective:

   To assess the reduction of microbial contamination (CFU/mL) on charcoal-infused toothbrushes compared to conventional toothbrushes after 21 days of use.

   Secondary Objective:

   To analyze potential oral health-based differences in microbial contamination
3. Study Design

   Type: Randomized Controlled Trial

   Design: Parallel, two-arm

   Duration: 21 days of intervention

   Randomization: 1:1 allocation (computer-generated random numbers)

   Blinding: Due to the visible color difference between charcoal-infused and conventional toothbrush bristles, participant blinding was not feasible.; laboratory analysis conducted under coded anonymity.

   Study Setting: Faculty of Dental Medicine, Rabat, Morocco
4. Study Population 4.1 Inclusion Criteria

   Dental students (4th or 5th year) aged 18-24 years.

   Regular manual toothbrush users.

   Good general and oral health.

   Willingness to comply with study instructions.

   Signed informed consent.

   4.2 Exclusion Criteria

   Irregular toothbrushing frequency.

   Refusal or allergy to charcoal products.

   Use of antiseptic toothpaste or mouthwash.

   Smoking or alcohol abuse.

   Systemic diseases or recent antibiotic therapy (<4 weeks).

   Plaque index >2 or gingival index >2.

   Periodontitis, orthodontic appliance wearers, or active oral infections.

   4.3 Sample Size

   A total of 32 participants (16 males, 16 females) were enrolled, divided equally between the two groups.
5. Study Procedures 5.1 Baseline Phase - Clinical Assessment

   Questionnaire: Participants completed an anonymous health and oral hygiene habits questionnaire (age, medical history, medication use, smoking, brushing frequency, and method).

   Clinical Examination: Using a mirror, dental explorer No. 23, and a periodontal probe, caries, restorations, and missing teeth were recorded using the DMF index.

   Plaque accumulation and gingival condition were assessed using the Silness & Löe plaque index and the Löe & Silness gingival index.

   5.2 Randomization and Group Allocation

   Eligible participants were randomly assigned to one of two groups:

   Group A: Colgate Double Action Medium toothbrushes with charcoal-infused bristles.

   Group B: Colgate Double Action Medium toothbrushes without charcoal. Both toothbrushes shared identical designs and bristle firmness.
6. Intervention Procedures 6.1 Participant Instructions

   Participants were instructed to:

   Brush twice daily for two minutes using the rolling technique.

   Use only the provided fluoride toothpaste (1450 ppm).

   Rinse the toothbrush with tap water only-without touching bristles.

   Avoid using any mouthwash or antiseptic toothpaste.

   Store the toothbrush vertically, bristles up, uncovered, at least 1-2 meters away from toilets.

   Record each brushing session on a standardized daily log sheet.

   Each participant received:

   One assigned toothbrush.

   One standardized toothpaste.

   One sterile storage pouch for post-study collection.
7. Sample Collection and Laboratory Procedures

   After 21 days, all used toothbrushes were collected in their sterile pouches and labeled with participant codes.

   7.1 Preparation of Blood Agar

   Columbia agar base was dissolved in distilled water according to manufacturer instructions, sterilized at 121°C for 15 minutes, and cooled to 45-50°C.

   Sterile defibrinated blood was aseptically added under a laminar flow hood.

   Approximately 20 mL of the medium was poured into sterile Petri dishes, solidified at room temperature, and stored inverted at 4°C until use.

   7.2 Preparation of Toothbrush Samples

   Approximately one-fourth of the bristles were aseptically cut with a sterile scalpel and transferred into sterile Petri dishes.

   The bristles were immersed in 5 mL of sterile saline solution for 10 seconds and vortexed to disperse microorganisms into suspension.

   7.3 Inoculation and Incubation

   A 200 µL aliquot of each suspension was inoculated on blood agar using sterile swabs.

   Plates were incubated at 37°C for 48 hours under aerobic conditions.

   7.4 Microbiological Analysis

   Colony-forming units (CFU) were manually counted using a digital colony counter.

   Results were expressed as CFU/mL.

   Statistical analyses were performed using Jamovi software.

   Shapiro-Wilk test for normality.

   Independent t-test or Mann-Whitney test for intergroup comparisons.

   Significance level set at p < 0.05.
8. Ethical Considerations

   The study protocol was approved by the Ethics Committee of the Faculty of Dental Medicine, Rabat.

   Written informed consent was obtained from all participants.

   Participant data were anonymized using unique codes.

   No personal identifiers were used in the analyses.

   The study involved minimal risk and no investigational drug or device.
9. Data Management and Confidentiality

   All data (clinical, microbiological, and questionnaires) were coded and stored securely. Only authorized investigators had access. Results were analyzed collectively, ensuring participant confidentiality.
10. Expected Outcomes

    The study is expected to demonstrate whether charcoal-impregnated bristle toothbrushes harbor fewer microorganisms after daily use, potentially supporting their antibacterial claims.
11. Study Limitations

    Convenience sampling limits external generalizability.

    Microbial identification limited to total CFU count without species differentiation.
12. Funding and Conflicts of Interest

No external funding or sponsorship was received. All materials were provided by the investigator. The authors declare no conflict of interest.

ELIGIBILITY:
Inclusion Criteria:

* Students of the Faculty of Dental Medicine of Rabat (4th or 5th year) aged 18-24 years.
* In good general health with no systemic diseases.
* Regular users of manual toothbrushes, brushing at least twice daily.
* Informed about the study and have signed informed consent.
* Willing to use the assigned toothbrush and follow study instructions for brushing technique, toothpaste use, and storage of the toothbrush.

Exclusion Criteria

* Irregular frequency of tooth brushing.
* Unwillingness to use a charcoal-impregnated toothbrush or known allergy to activated charcoal.
* Use of antiseptic mouthwash and/or antiseptic toothpaste.
* Smoking.
* Presence of systemic disease.
* Current or recent antibiotic therapy (within the 4 weeks prior to the study).
* High plaque index (>2, Silness & Löe).
* Periodontitis.
* Severe gingivitis (gingival index >2, Löe & Silness).
* Wearing orthodontic appliances.
* Current oro-pharyngeal infections.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Reduction of microbial contamination on toothbrush bristles | 21 days
  The primary outcome is the number of colony-forming units (CFU/mL) measured on toothbrush bristles after 21 days of use. A quarter of the bristles from each brush is cut and placed in sterile saline, vortexed to create a suspension, and 200 µL is inoculated on blood agar plates. Plates are incubated at 37°C for 48 hours, and CFU are counted manually. This outcome assesses the effectiveness of charcoal-impregnated bristles in reducing microbial contamination compared to conventional toothbrushes.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine of Rabat, Mohammed V University, Rabat, Al Irfane, Morocco